CLINICAL TRIAL: NCT02264288
Title: A Phase 2 Multicenter, Randomized, Doubleblind, Placebo-Controlled, Dose Range Finding Study to Evaluate the Efficacy and Safety of Intramuscular Injection of Human Placenta-derived Cells (Pda-002) in Subjects Who Have Diabetic Foot Ulcer With Peripheral Arterial Disease
Brief Title: Efficacy and Safety of Intramuscular PDA-002 in Subjects Who Have Diabetic Foot Ulcer With and Without Peripheral Arterial Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision with all subjects completing at least 1 year follow-up
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-PDA-002-DFU-002
Record Dates: First submitted 2014-10-02; First posted 2014-10-15 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Arterial Disease; Diabetic Foot
Keywords: Peripheral Arterial Disease; Diabetic Foot
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 x 10^6 cells (Experimental): Human Placenta Derived cells (PDA-002) administered intramuscularly (IM) on Study Days 1 and 8
  Interventions: Biological: 3 x 10^6 cells
- 10 x 10^6 cells (Experimental): 10 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 10 x 10^6 cells
- 30 x 10^6 cells (Experimental): 30 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 30 x 10^6 cells
- Placebo (Placebo Comparator): Identically matching placebo administered IM on Study Days 1 and 8
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: 3 x 10^6 cells — 3 x 10^6 cells administered on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 3 x 10^6 cells
Biological: 10 x 10^6 cells — 10 x 10^6 Human Placenta Derived cells (PDA-002) administered on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 10 x 10^6 cells
Biological: 30 x 10^6 cells — 30 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 30 x 10^6 cells
Other: Placebo — Identical matching placebo administered IM on Study Days 1 and 8
  Arms: Placebo

SUMMARY:
The PDA-002-DFU-002 trial is a Phase 2, multicenter, randomized, double blind, placebo controlled, dose range finding study. The study will enroll approximately 133 subjects in four treatment groups. The primary objective of the study is to assess the efficacy and safety of PDA-002 administered intramuscular (IM) in subjects who have DFU with and without PAD. The secondary objective is to explore potential clinical efficacy by assessing changes in vascular parameters such as Ankle-Brachial Index and Toe-Brachial Index (ABI and/or TBI), Transcutaneous oxygen measurements (TcPO2).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, at least 18 years of age or older at the time of signing the informed consent document.
2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Diabetes mellitus Type 1 or Type 2.
5. Diabetic foot ulcer with severity of Grade 1 (full thickness only) or Grade 2 on the Wagner Grading Scale (Appendix A) of greater than one month duration which has not adequately responded to conventional ulcer therapy with a size of at least of 1cm2 except if present on the toe. The maximum lesion size range in the index ulcer is ≤ 10cm2. The measurement of the index ulcer is to be evaluated and measured after debridement (if necessary) at the Screening Visit. If located on the plantar aspect of the foot, the index ulcer must be able to be adequately offloaded in the assessment of the investigator.
6. No planned revascularization or amputation over the next 3 months after Screening visit, in the opinion of the Investigator.
7. Screening should not begin until at least 14 days after a failed reperfusion intervention and at least 30 days after a successful reperfusion intervention.
8. Subjects should be receiving appropriate medical therapy for hypertension and diabetes any other chronic medical conditions for which they require ongoing care.
9. A female of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test prior to treatment with study therapy. In addition, sexually active FCBP must agree to use 2 of the following adequate forms of contraception methods simultaneously such as: oral, injectable, or implantable hormonal contraception; tubal ligation; IUD; barrier contraceptive with spermicide or vasectomized partner for the duration of the study and the Follow-up Period.
10. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP for the duration of the study and the Follow-up Period.

Exclusion Criteria:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he or she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Pregnant or lactating females.
5. Subjects with a body mass index > 45 kg/m2 at Screening.
6. AST (SGOT) or ALT (SGPT) > 2.5 x the upper limit of normal (ULN) at Screening.
7. Patient on renal dialysis for abnormal kidney function.
8. An ABI < 0.4 and or TBI < 0.3 in the leg with the index ulcer.
9. Bilirubin level > 2 mg/dL (unless subject has known Gilbert's disease) at Screening.
10. Untreated chronic infection or treatment of any infection with systemic antibiotics, including the ulcer site, must be free of antibiotics within 1 week prior to dosing with IP.
11. Active osteomyelitis, infection, or cellulites at or adjacent to the index ulcer. Patients with a history of being treated for an osteomyelitis without a surgical resection.
12. Index ulcer that has decreased or increased in size by ≥ 30% during the Screening/Run-In/ Pre-Treatment Period.
13. Active Charcot Neuroarthropathy in the foot with the index ulcer
14. Pain at rest due to limb ischemia.
15. Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 180 mmHg during Screening at 2 independent measurements taken while subject is sitting and resting for at least 5 minutes).
16. Poorly controlled diabetes mellitus (hemoglobin A1c > 12% or a screening serum glucose of ≥ 300mg/dl).
17. Untreated proliferative retinopathy.
18. History of malignant ventricular arrhythmia, CCS Class III-IV angina pectoris, myocardial infarction/ percutaneous coronary intervention (PCI) / coronary artery bypass graft (CABG) in the preceding 6 months prior to signing the informed consent form (ICF), pending coronary revascularization in the following 3 months, transient ischemic attack/cerebrovascular accident in the preceding 6 months, prior to signing the ICF, and/or New York Heart Association [NYHA] Stage III or IV congestive heart failure.
19. Abnormal ECG: new right bundle branch block (BBB) ≥ 120 msec in the preceding 3 months prior to signing the ICF.
20. Uncontrolled hypercoagulation syndrome.
21. Life expectancy less than at 2 years at the time of signing the ICF due to concomitant illnesses.
22. In the opinion of the Investigator, the subject is unsuitable for cellular therapy.
23. History of malignancy within 5 years prior to signing the ICF except basal cell or squamous cell carcinoma of the skin or remote history of cancer now considered cured or positive Pap smear with subsequent negative follow-up.
24. History of hypersensitivity to any of the components of the product formulation (including bovine or porcine products, dextran 40, and dimethyl sulfoxide [DMSO]).
25. Subject has received an investigational agent -an agent or device not approved by the US Food and Drug Administration (FDA) for marketed use in any indication- within 90 days (or 5 half-lives, whichever is longer) prior to treatment with study therapy or planned participation in another therapeutic study prior to the completion of this study.
26. Subject has received previous investigational gene or cell therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2014-10-23 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Complete wound closure of the index ulcer | Up to 4 months
  Complete wound closure is defined as closure of the index ulcer and retaining wound closure for the subsequent 4 weeks
Safety (adverse events [type, frequency, and severity of AEs, and relationship of AEs to study drug], laboratory abnormalities, and hospitalizations | Up to 24 months
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study.

SECONDARY OUTCOMES:
Time to ulcer closure | Up to 6 months
  The time period for the index ulcer to close
Ankle Brachial Index (ABI ) and Toe-Brachial Index (TBI) | Up to 6 months
  ABI and TBI will be calculated by dividing the systolic blood pressure at the ankle or toe by the systolic blood pressures (Doppler technique) in the arm
50% Closure of Index Ulcer | Up to 24 months
  The proportion of subjects with at least 50% closure of the index ulcer
Transcutaneous oxygen | Up to 6 months
  Transcutaneous oxygen measurements determine the oxygen level in tissue below the skin
Time to amputation, ulcer opening closing, gangrene and infection | Up to 24 months
  Time to major amputation (above the ankle) of treated leg, minor amputations, to re-opening of ulcer, time to doubling / halving of index ulcer total surface area from baseline, de novo gangrene and foot wound infection
Wagner Grading Scale | Up to 24 months
  The Wagner system assesses ulcer depth and the presence of osteomyelitis or gangrene by using the following grades: grade 0 (pre-or postulcerative lesion), grade 1 (partial/full thickness ulcer), grade 2 (probing to tendon or capsule), grade 3 (deep with osteitis), grade 4 (partial foot gangrene), and grade 5 (whole foot gangrene).
Rutherford Criteria | Up to 6 months
  The Rutherford classification is a clinical staging system for describing peripheral arterial disease.
36-item Short Form Health Survey (SF-36) | Up to 6 months
  A validated measurement of health related quality of life
Diabetic Foot Ulcer Scale Short Form (DFS-SF) index ulcer | Up to 6 months
  A measurement of the impact of diabetic foot ulcer on a patient's quality of life.
Patient Global Impression of Change in Neuropathy (PGICN) | Up to 24 months
  Assessment of changes in neuropathy over time
European Quality of Life: EuroQOL-5D- health utility index assessment (EQ-5D) | Up to 6 months
  A standardized instrument used as a measure of health outcome
Number of all ulcers | Up to 24 months
  The total number of ulcers
Leg rest pain score | Up to 24 months
  A visual analog scale (VAS) graded from 0 (pain free) to Grade 10 (maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Solveig Ericson, MD, Study Director — Celularity Incorporated
Locations (55):
- United States (55):
  - Cardiology PC, Birmingham, Alabama
  - TFi Medical, Mobile, Alabama
  - East Valley Foot and Ankle Specialist, Mesa, Arizona
  - Carl T. Hayden Veterans Affairs Medical Center, Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Aung Foothealth Clinics and Advanced Wound Care Center, Tucson, Arizona
  - Northeast Arkansas Baptist Clinic, Jonesboro, Arkansas
  - Jeffrey A Klemes DPM, Beverly Hills, California
  - Center for Clinical Research Inc., Castro Valley, California
  - Reliance Clinical Research, Chino, California
  - Limb Preservation Platform, INC., Fresno, California
  - Foot and Ankle Clinic, Los Angeles, California
  - UCLA, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Stanford, California
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Barry University, Fort Lauderdale, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - The Research Center, Hialeah, Florida
  - University of Florida, Jacksonville, Florida
  - Solutions Through Advanced Research Inc., Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Well Pharma Medical Research Corporation, Miami, Florida
  - GF Professional Research Group Corporation, Miami Lakes, Florida
  - Med-Care Research Inc, North Miami Beach, Florida
  - Podiatry 1st, Belleville, Illinois
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Weill Foot & Ankle Institute, Des Plaines, Illinois
  - Rosalind Franklin University of Medicine and Science, North Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Foot and Ankle Center of Illinois, Springfield, Illinois
  - CGH Medical Center Main Clinic, Sterling, Illinois
  - Hamilton Foot Care, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Northwest Hospital, Randallstown, Maryland
  - Revive Research Institute, Sterling Heights, Michigan
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Office of Michael J. De Marco, DPM, Tinton Falls, New Jersey
  - Ocean City Foot and Ankle Assoc, Toms River, New Jersey
  - Animas Foot and Ankle, Gallup, New Mexico
  - Office of Gerard J. Furst, DPM, PLLC, East Setauket, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - UNC Hospitals University of North Carolina, Chapel Hill, North Carolina
  - Clinical Research Associates of Central Pennsylvania, Duncansville, Pennsylvania
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Premier Vein and Vascular Center, Houston, Texas
  - Complete Family Foot Care - McAllen Office, McAllen, Texas
  - Endeavor Clinical Trials PA, San Antonio, Texas
  - SAM Clinical Research Center, San Antonio, Texas
  - Advanced Foot & Ankle Center, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
  - 1Foot 2Foot Centre for Foot & Ankle Care PC, Suffolk, Virginia
  - Milwaukee Foot & Ankle Specialists, Wauwatosa, Wisconsin